CLINICAL TRIAL: NCT02737488
Title: Helping Children With Trauma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-01251
Record Dates: First submitted 2016-04-08; First posted 2016-04-14 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Trauma; Post-Traumatic Stress Disorder
Keywords: Therapy; Trauma Systems Therapy
MeSH Terms: conditions — Wounds and Injuries; Stress Disorders, Post-Traumatic | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TST (Experimental)
  Interventions: Behavioral: Trauma Systems Therapy (TST)
- TAU Group (Active Comparator)
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Trauma Systems Therapy (TST) — Treatment will be delivered by clinicians and trainees working at the CSC who have been trained in delivering TST. Participants who begin treatment in the safety-focused phase will have their treatment sessions in their homes. Whenever a child enters a different phase of treatment, he or she will go to the site for office visits. At the beginning of treatment, TST clinicians will do a brief diagnostic assessment. All documentation that is completed by the clinician as part of TST treatment at the NYU Langone Medical Center will be documented using Epic, a standard of care integrated health information system for patient safety. Although we are not providing the CSC's standard of care in this study,we are replicating standard care as TST is standard care in other settings. Providing medication is part of standard TST treatment and conforms to good usual practice integrated with psychotherapy. Medication will not be prescribed for research purposes.
  Arms: TST
Behavioral: Treatment as Usual (TAU) — Youth in the control group will be referred to a mental health clinic in close proximity to their residence, in order to receive an evaluation and trauma treatment as usually provided. It cannot be specifically determined, in advance, the nature of this treatment.
  The clinics will be contacted after the family enrolls to determine if there was a specific protocol followed. An NYU CSC research coordinator will contact the clinic and assist in scheduling the subject's first visit. Families who do not enroll in any community treatment or dropout of treatment will be followed according to the research protocol for data collection. At the 3, 6, and 9 month assessments, the research coordinator will request the patient's records from the community treatment clinic they are attending in order to track and keep record of the youth's treatment modality, progress, and visit frequency.
  Arms: TAU Group

SUMMARY:
The purpose of this study is to evaluate if a trauma treatment called Trauma Systems Therapy (TST) decreases children's mental health symptoms (such as acting out, not controlling their emotions, etc.) as a result of a traumatic event (or events). A traumatic event or events can include experiencing or witnessing violence, excessive bullying, war, car accident, serious injury, getting mistreated or anything else that makes one feel scared or frightened. Children/teens who experience traumatic events have been shown to be at higher risk of poor mental and physical health. Trauma can impact family life, school life and interpersonal relationships well into adulthood. Unfortunately, most children who have experienced traumatic events do not undergo treatment. Although promising treatments do exist, most do not address the complexity of trauma, particularly related to ongoing stress and threats to safety in their environments. One hundred and twenty eligible youth will be randomized to receive either treatment with TST at NYU's Child Study Center or trauma treatment as usual (TAU) at a community mental health clinic.

It is hypothesized that:

* Youth receiving TST will demonstrate a greater decrease in Post-Traumatic Stress Disorder (PTSD) symptoms at the 3, 6, and 9-month follow-up assessments compared to youth receiving treatment as usual (TAU) in the community.
* Youth receiving TST will demonstrate a greater decrease in symptoms of depression, anxiety and problem behaviors (aggression, violence, self-destructive behaviors, etc.) at the 3-, 6- and 9-month follow-up assessments compared to youth receiving TAU.
* Youth receiving TST will have fewer acute mental health service events, such as psychiatric hospitalizations and ED visits compared to youth receiving TAU.
* Greater fidelity to the TST model is associated with better treatment outcomes among youth receiving TST.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 7 and 17.
* Have experienced a trauma and have symptoms of that trauma for more than 1 month
* Have a legal guardian who is willing to give consent and a primary caregiver who will be available for assessments.

Exclusion Criteria:

* Reside outside the study area
* Currently participating in another study
* Do not speak English
* Receive psychotherapy elsewhere
* Have a sibling already participating in the study
* Are acutely suicidal or homicidal
* Demonstrate they are in immediate danger
* Legal guardian does not give consent
* If the primary caregiver does not speak English, does not have consistent access to a telephone, does not have the capacity to answer questions, the child will be excluded.
* If a potential subject has started, stopped, or changed a psychotropic medication within 2 weeks of their intake appointment. If the family is willing to wait for 2 weeks the participant may then be eligible.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2016-02-01; Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
UCLA-Post Traumatic Stress Disorder-Reaction Index-DSM-IV (UCLA-PTSD-RI-DSM-IV) | 9 Months
  The primary outcome (PTSD symptom severity) will be collected at 3, 6 and 9 months post-randomization in addition to baseline. The effect of TST compared with TAU will be evaluated based on mixed effects model for longitudinal data.
Child Stress Disorder Checklist (CSDC) | 9 months
  The primary outcome (PTSD symptom severity) will be collected at 3, 6 and 9 months post-randomization in addition to baseline. The effect of TST compared with TAU will be evaluated based on mixed effects model for longitudinal data.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Saxe, MD, Principal Investigator — Glenn.Saxe@nyumc.org
Locations (1):
- NYU Langone Medical Center, New York, New York, United States